CLINICAL TRIAL: NCT07018973
Title: The Role of Generative Artificial Intelligence Supported Morphological Analysis on Problem Solving Skills and Creative Thinking Disposition of Nursing Students: A Randomized Controlled Trial
Brief Title: The Effect of Artificial Intelligence Supported Morphological Analysis on Problem Solving and Creative Thinking Disposition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Nurcan Çalışkan, Prof, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025-616
Record Dates: First submitted 2025-05-29; First posted 2025-06-13 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Generative Artificial Intelligence; Creative Thinking; Problem Solving; Morphological Analysis and Classification; Nursing; Student
Keywords: Creative Thinking; Problem Solving; Morphological Analysis; Nursing; Student; Generative Artificial Intelligence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GAISMA (Experimental)
  Interventions: Other: GAISMA
- Control (Other)
  Interventions: Other: Control

INTERVENTIONS:
Other: GAISMA — After the pre-test and randomization, the experimental group will first start the morphological analysis application. After completing a certain period of time, copies of the matrix and suggestion studies will be taken and they will be allowed to use the generative artificial intelligence application. At the end of the application, a post-test will be applied. In addition, an opinion form will be given and their opinions about the morphological analysis method, the use of generative artificial intelligence and the use of artificial intelligence with the morphological analysis method and how it affects them will be taken.
  Arms: GAISMA
Other: Control — In the control group, morphological analysis will be applied. Post-tests will be applied at the end of the application. Finally, their opinions about the morphological analysis method and how it affects them will be taken by giving an opinion form.
  Arms: Control

SUMMARY:
It will be conducted as a two-group, pretest-posttest, randomized controlled study to determine the effect of generative artificial intelligence-supported morphological analysis on nursing students' problem solving skills and creative thinking tendencies. This study will be conducted with third year students who enrolled in Gazi University Faculty of Health Sciences, Department of Nursing, HEM 312 Critical Thinking in Nursing course for the first time in the spring semester of the 2024-2025 academic year and agreed to participate in the study. Data will be collected using the "Inclusion Form", "Descriptive Characteristics Form", "Marmara Creative Thinking Dispositions Scale", "Problem Solving Skills Scale for Adults" and "Morphological Analysis and Generative Artificial Intelligence Application Opinion Form". Students who meet the inclusion criteria will be randomized into intervention and control groups according to the midterm exam results of the course. At the end of the intervention, post-tests (Marmara Creative Thinking Dispositions Scale and Problem Solving Skills Scale for Adults) will be administered. The control group will be allowed to use the generative artificial intelligence after completing the post-tests. When the application is completed, students will be given an opinion form and their opinions will be taken. The data of the intervention and control groups will be analyzed with SPSS in computer environment.

DETAILED DESCRIPTION:
Students assigned to groups will start morphological analysis for the problems to be given within the scope of patient safety objectives in groups of 5-6 people. One group in the experimental and one group in the control group will be distributed in such a way that the same problem will coincide. Information about the morphological analysis method will be given before the application. The matrix papers made in morphological analysis will be distributed to the groups and the students will be enabled to create their matrices, select their combinations and produce solutions. Researchers will provide coordination in groups. One of the researchers took a course on creative thinking techniques. After the application, the study will be completed with the presentation of matrix, combination and solution proposals of the experimental and control groups. Thus, the implementation will be completed in one day and the study will be finalized by taking post-tests and opinion forms.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Taking HEM 312 Critical Thinking in Nursing course for the first time

Exclusion Criteria:

* Not attending more than 30% of HEM 312 Critical Thinking in Nursing course
* To have received a training on Morphological Analysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2025-06-12 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Marmara Creative Thinking Dispositions Scale | Baseline and within 24 hours after intervention
  The scale, which is suitable for use on adults, consists of 25 items and 6 dimensions. The sub-dimensions are named as innovation seeking, courage, self-discipline, curiosity, doubt and flexibility. The five-point Likert-type scale consists of options as 1 - never, 2 - rarely, 3 - occasionally, 4 - usually and 5 - always. The scale explains 55.904% of the total variance. Cronbach's alpha internal consistency coefficient for the whole scale was calculated as 0.87. There are no reverse items in the scale. The high score obtained from each sub-dimension of the scale indicates that the individual has the characteristic evaluated by the relevant sub-dimension. The scale also gives a total creative thinking tendencies score. When scoring the scale, the average of the sub-dimensions and the total score are taken.
Problem Solving Skills Scale for Adults | Baseline and within 24 hours after intervention
  The scale was administered to 550 adults to assess their problem solving skills for various problems in their daily lives and Cronbach's Alpha internal consistency coefficient was found to be 0.88. The scale is a Likert-type scale consisting of 18 items scored between 1-5. The options in the scale are 1-Never, 2-Rarely, 3-Sometimes, 4-Frequently, 5-Always. As a result of the factor analysis, the scale consists of 5 factors: "Thinking about the Effects of Solving the Problem" (5 items), "Problem Solving through Modeling" (3 items), "Searching for Alternative Solutions" (3 items), "Determination in Applying the Determined Solution" (3 items), "Analyzing the Problem Encountered" (3 items). There are no reverse items in the scale. In addition, the lowest score is 18 and the highest score is 90. The high score obtained from each sub-dimension of the scale indicates that the individual has the characteristic evaluated by the relevant sub-dimension.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Nursing, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No